CLINICAL TRIAL: NCT05026853
Title: Patient-Reported Outcomes Measurement Information System Integration Into Rheumatology Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Frederick G L Huetwell Professor of Rheumatology and Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00149448; K24AR063120 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Rheumatic Diseases
Keywords: Health-related quality of life; PROMIS
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: There will be two arms (1: 1 randomization) of the trial to assess PRO integration into care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO Integration into Clinical Practice (Experimental): PRO scores will be shared with patients and healthcare providers (HCPs) via an emailed report card
  Interventions: Behavioral: PRO Integration into Clinical Practice
- Usual Care (No Intervention): Patients and HCPs will not receive an emailed PROMIS score report. PROMIS scores, however, will be available in the EMR as usual.

INTERVENTIONS:
Behavioral: PRO Integration into Clinical Practice — HCPs will document their discussion and recommendations/referrals in MiChart (Epic EMR)
  Arms: PRO Integration into Clinical Practice

SUMMARY:
This study will examine the impact of providing patient-reported outcomes measurement information system (PROMIS) scores to patients before appointments with their healthcare provider.

ELIGIBILITY:
Inclusion Criteria for patients:

* New and established patients seeking care at Michigan Medicine rheumatology clinics
* Patients should have access to the patient portal in MiChart patient portal
* Patients should have access to the internet at home to be able to complete the PROMIS PRO measures and study surveys online
* Patients should have completed PROMIS pain, physical function, and sleep disturbance measures at least one day before their baseline appointment
* At least one of the PROMIS PRO scores should be in the concerning zone (pain intensity ≥ 5, physical function ≤ 40, or sleep disturbance ≥ 60).

Exclusion Criteria:

* Non-English speakers
* under 18 years of age

Inclusion Criteria for providers:

* Rheumatology health care providers, including clinicians and advanced practice providers at Michigan Medicine who are currently treating rheumatology patients

Exclusion Criteria:

* Those not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gedert R, Ochocki D, Kortam N, Huang S, Nagaraja V, Chakrabarti K, Ford J, Garber M, Lee J, Ognenovski V, Roofeh D, Cella D, Khanna D. A pilot trial of integrating the Patient-Reported Outcome Measurement Information System (PROMIS(R)) into rheumatology care. Clin Exp Rheumatol. 2025 Jan;43(1):112-118. doi: 10.55563/clinexprheumatol/fp914f. Epub 2024 Oct 25. PMID 39480493

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
Started | 55 | 55
Week 2 Follow-up | 35 | 45
Week 12 Follow-up | 30 | 39
Completed | 30 | 39
Not Completed | 25 | 16
Not completed — Cancelled appointment | 1 | 0
Not completed — Excluded due to technical difficulties with generating scorecard | 8 | 0
Not completed — Did not complete 12-week survey | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO Integration Into Clinical Practice | Usual Care | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 39 | 86
  >=65 years | 8 | 16 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.9) | 55.2 (14.3) | 53.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 46 | 49 | 95
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 53 | 51 | 104
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 55 | 110
PROMIS Domain Scores [Mean (Standard Deviation); unit: score] — Pain intensity is reported as a scaled score of 0-10, where 0 indicates no pain and 10 indicates worst possible pain. The scores in PROMIS measures are computed to a T-score metric, where 50 represents the mean for US general population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measured, except physical function where a lower T-score indicates increased impairment. With physical function, a higher score indicates greater function and with sleep disturbance, a lower score indicates less disturbance.
  score
    Pain Intensity, 0-10 scale, where 0 is no pain and 10 is worst possible pain | 5.2 (1.8) | 5.5 (2.1) | 5.3 (1.9)
    Physical Function, T-score. A higher score indicates greater function. | 38.2 (7.0) | 37.7 (6.3) | 37.9 (6.6)
    Sleep Disturbance, T-score. A lower score indicates less disturbance. | 58.2 (7.4) | 57.1 (9.2) | 57.6 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Appointments at Which Patient-Reported Outcomes Measurement Information System (PROMIS) Scores Are Documented in the Electronic Medical Record (EMR) Note by the Participating Health Care Provider (HCP)
Description: Documentation in EMR notes will be categorized as either 'yes' or 'no' and identified through EMR data pulls. Percent of appointments is shown by the count (and percentage) of participants for whom PROMIS scores were documented in the EMR for their appointment.
Time Frame: Up to 3 months
Population: 1 appointment was cancelled and 8 were unable to receive score card due to technical difficulties.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
Number analyzed (Participants) | 46 | 55
Participants | 23 | 7

2. Secondary Outcome: Percent of Appointments at Which Referrals/Recommendations Related to PROMIS Scores Are Documented in the EMR Note by the Participating HCP
Description: Documentation in EMR notes will be either 'yes' or 'no' and identified through EMR data pulls. Percent of appointments is shown by the count (and percentage) of participants for whom referrals were documented in the EMR.
Time Frame: Up to 3 months
Population: 1 appointment was cancelled and 8 were unable to receive score card due to technical difficulties.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
Number analyzed (Participants) | 46 | 55
Participants | 17 | 6

3. Secondary Outcome: Quality of Patient-provider Communication
Description: Patient-provider communication is measured using the Interpersonal Processes of Care (IPC) Survey (29 items), which measures 7 subscales. For the subscales "elicited concerns/responded", "explained results/medications", "patient-centered decision making", and "compassionate, respectful" a higher score is better. For the subscales "hurried communication", "discrimination", and "disrespectful office staff" a lower score is better. (score for each subscale ranges from 1-5; + indicates a higher score is better, - indicates a lower score is better). Questions were not mandatory.
Time Frame: Up to 2 weeks
Population: Not all subjects completed every question. Some subjects skipped questions. In the usual care arm, no question was answered by more than 43 people.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
Number analyzed (Participants) | 35 | 43
score on a scale
  Communication: Hurried communication (-) | 1.3 (0.5) | 1.2 (0.5)
  Communication: Elicited concerns, responded (+) | 4.1 (1.3) | 4.5 (1.0)
  Communication: Explained results, medications (+): number analyzed (Participants) | 34 | 43
  Communication: Explained results, medications (+) | 4.0 (1.2) | 4.0 (1.1)
  Decision making: Patient-centered decision (+): number analyzed (Participants) | 35 | 42
  Decision making: Patient-centered decision (+) | 4.0 (1.3) | 4.0 (1.3)
  Interpersonal style: Compassionate, respectful (+): number analyzed (Participants) | 34 | 42
  Interpersonal style: Compassionate, respectful (+) | 4.4 (1.0) | 4.5 (0.9)
  Interpersonal style: Discrimination (-): number analyzed (Participants) | 34 | 42
  Interpersonal style: Discrimination (-) | 1.1 (0.4) | 1.0 (0.2)
  Interpersonal style: Disrespectful office staff (-): number analyzed (Participants) | 33 | 41
  Interpersonal style: Disrespectful office staff (-) | 1.0 (0.0) | 1.0 (0.2)

4. Secondary Outcome: Change in Score of the Most Bothersome PROMIS Domain
Description: Change in score of PROMIS domain deemed most bothersome by each subject at baseline. Pain intensity is reported as a scaled score of 0-10, where 0 is no pain and 10 is the worst pain possible. Physical function and sleep disturbance are reported as T-scores.
  The scores in PROMIS measures are computed to a T-score metric, where 50 represents the mean for US general population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measured, except physical function where a lower T-score indicates increased impairment. With physical function, a higher score indicates greater function and with sleep disturbance, a lower score indicates less disturbance.
Time Frame: Baseline, 3 months
Population: The most concerning domain for subjects in each arm was analyzed.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
Number analyzed (Participants) | 29 | 39
score
  Pain Intensity, 0-10 scale: number analyzed (Participants) | 7 | 14
  Pain Intensity, 0-10 scale | -1.1 (2.5) | -0.9 (2.4)
  Physical Function, T-score. A higher score indicates higher function.: number analyzed (Participants) | 14 | 19
  Physical Function, T-score. A higher score indicates higher function. | -0.5 (2.6) | 1.1 (4.8)
  Sleep Disturbance, T-score. A lower score indicates less disturbance.: number analyzed (Participants) | 8 | 6
  Sleep Disturbance, T-score. A lower score indicates less disturbance. | -2.8 (6.6) | -3.3 (6.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | PRO Integration Into Clinical Practice | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT05026853/Prot_SAP_000.pdf